CLINICAL TRIAL: NCT02874898
Title: Marijuana Use, Extinction Learning, and Exposure Therapy in Individuals With PTSD
Brief Title: Short-Term Exposure for PTSD
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michele Bedard-Gilligan, Assistant Professor, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001289; 1R34DA040034-01A1 (NIH)
Record Dates: First submitted 2016-08-16; First posted 2016-08-22 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Chronic Post-Traumatic Stress Disorder; Marijuana Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy marijuana use (Active Comparator): Heavy marijuana users with PTSD
  Interventions: Behavioral: Brief Imaginal Exposure
- No marijuana use (Active Comparator): Non-marijuana users with PTSD
  Interventions: Behavioral: Brief Imaginal Exposure

INTERVENTIONS:
Behavioral: Brief Imaginal Exposure — Psychoeducation and imaginal exposure components of full prolonged exposure, in which patients relive the trauma vividly and process thoughts and feelings related to it

SUMMARY:
This study examines how marijuana use affects processes related to recovery from chronic posttraumatic stress disorder (PTSD). Half the participants will be individuals with chronic PTSD and heavy marijuana use and half will be individuals with chronic PTSD and no marijuana use. This study will assess how individuals with PTSD with heavy or no marijuana use perform on a discriminative conditioning and extinction paradigm designed to measure fear extinction learning, and how they respond to a brief daily imaginal exposure treatment in regards to PTSD symptom reduction.

DETAILED DESCRIPTION:
In this study, 36 patients with chronic PTSD and heavy marijuana use (heavy) and 36 patients with chronic PTSD and no marijuana use (no use) will be recruited to examine the effects of marijuana use on behavioral (emotional experiencing), physiological (skin conductance, acoustic startle) and biological (cortisol, blood pressure) responding on a well-established discriminative conditioning and extinction paradigm. To examine real world therapeutic implications, we will also examine how individuals with PTSD and heavy or no marijuana use differentially respond to a brief (6 session, 50 min) daily imaginal exposure (IE) treatment. Throughout treatment, we will monitor level of cannabis metabolites in urine samples of marijuana users to correlate effects to outcomes and preliminarily explore how varying levels of cannabis metabolites affect extinction processes. Independent evaluators will assess patients at baseline, 4 weeks, and 12 weeks following study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Current PTSD diagnosis based on DSM-5 criteria, with a minimum duration of 12 weeks since the traumatic event;
2. Between the age of 18 and 65;
3. Current heavy marijuana use (5+ days per week for 3+ months) or no marijuana use in the last 3 months
4. Current diagnosis of a cannabis use disorder based on DSM-5 or no current diagnosis of a substance use disorder

Exclusion Criteria:

1. Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by the DSM-5.
2. Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
3. Unwilling or unable to discontinue current trauma-focused psychotherapy
4. Any previous experience with prolonged exposure (PE) treatment
5. No clear trauma memory or trauma before age 3
6. Unstable dose of psychotropic medications in the prior 3 months
7. Ongoing intimate relationship with the perpetrator (in assault related PTSD cases).
8. Current diagnosis of a substance use disorder according to DSM-5, other than marijuana in the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Symptom Scale- Interview Version (PSS-I) | 12 Weeks
  The PSS-I assesses symptoms of PTSD as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) and is administered at baseline, 4 week, and 12 week follow up to assess change in PTSD symptoms
Treatment drop-out | 2 Weeks
  Defined as completion of less than 5 of 6 sessions of IE treatment

SECONDARY OUTCOMES:
Change in Quick Inventory of Depressive Symptomatology (QIDS-SR16) | baseline, 4 week, and 12 Weeks
  The QIDS-SR16 assesses symptoms of depression as defined by the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) and is administered at baseline, 4 week, and 12 week follow up to assess change in depression symptoms.
Change in Marijuana Problems Scale (MPS) | baseline, 4 week, and 12 Weeks
  The MPS is a self-report that assesses the impacts of marijuana on various areas of life, including motivation and productivity, social relationships, work and finances, self-esteem, memory impairment, legal problems, and physical health. The MPS is administered at baseline, 4 week and 12 week follow up to assess change in marijuana abuse.
Change in Marijuana Frequency and Quantity | baseline, 4 week, and 12 Weeks
  The Marijuana Frequency and Quantity Scale assesses the frequency and quantity of marijuana use and is administered at baseline, 4 week and 12 week follow up to assess changes in marijuana use.

CONTACTS AND LOCATIONS:
Overall Officials: Michele A Bedard-Gilligan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No